CLINICAL TRIAL: NCT01817738
Title: A Randomised, Double-blind, Placebo-controlled, Phase I/II Trial of RNActive®-Derived Cancer Vaccine (CV9104) in Asymptomatic or Minimally Symptomatic Patients With Metastatic Castrate-refractory Prostate Cancer
Brief Title: Trial of RNActive®-Derived Prostate Cancer Vaccine in Metastatic Castrate-refractory Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Follow up period after primary analysis was prematurely stopped because more mature data will not impact the study outcome
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV-9104-004
Record Dates: First submitted 2013-02-08; First posted 2013-03-25 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Castrate-refractory
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CV9104 (Active Comparator): CV9104 intradermal injection
  Interventions: Biological: CV9104
- Placebo (Placebo Comparator): Placebo intradermal injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CV9104 — Intradermal injection of CV9104
  Arms: CV9104
Biological: Placebo — Intradermal injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the new RNActive®-derived prostate cancer vaccine CV9104 prolongs survival in patients with asymptomatic or minimally symptomatic metastatic prostate cancer that is castrate resistant.

DETAILED DESCRIPTION:
The study is the first clinical study with the new prostate cancer vaccine CV9104. This vaccine is composed of 6RNActive®-based compounds, each encoding for an antigen that is overexpressed in prostate cancer compared to healthy tissues. RNActive®-based vaccines are a novel class of vaccines based on messenger RNA.

The study is a double-blind randomized placebo-controlled phase I/II trial in men with asymptomatic- minimally symptomatic metastatic castrate-refractory prostate cancer.

The phase 1 (safety lead- in) part of the trial has the primary objective to assess the safety of CV9104 and to determine the dose for the randomized phase II part.

The primary objective of the phase II part is to compare overall survival in patients treated with CV9104 compared to patients treated with placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male, age ≥18 years
2. Histologically confirmed castrate refractory metastatic adenocarcinoma of the prostate with progressive disease after surgical castration or during androgen suppression therapy including a GNRH agonist or antagonist and after at least 1 additional anti-hormonal manipulation; and serum testosterone level of < 50 ng/dL or < 1.7 nmol/L

   Progression will be confirmed either
   * radiologically or
   * by 2 consecutive rises of PSA, measured at least 1 week apart, resulting at least in a 50% increase over the nadir and a PSA > 2 ng/mL.
   * An antiandrogen withdrawal response must have been excluded after discontinuation of antiandrogen therapy for at least 6 weeks.
3. Metastatic disease confirmed by imaging
4. ECOG performance status 0 or 1

Key Exclusion Criteria:

1. Previous immunotherapy for PCA (e.g. sipuleucel-T [Provenge®], experimental cancer vaccines or ipilimumab [Yervoy®]).
2. Treatment with any investigational anticancer agents within 4 weeks prior to first dose of study drug
3. Systemic treatment with immunosuppressive agents
4. Active skin disease (atopic eczema, psoriasis) in the areas for vaccine injection (upper arms or thighs) preventing the administration of i.d. injections into areas of healthy skin.
5. History of or current autoimmune disorders
6. Primary or secondary immune deficiency.
7. Seropositive for human immunodeficiency virus, hepatitis B virus (except after hepatitis B vaccination) or hepatitis C virus infection.
8. Symptomatic congestive heart failure (New York Heart Association 3 or 4), unstable angina pectoris or myocardial infarction, significant cardiac arrhythmia, history of stroke or transient ischemic attack, all within 6 months prior to enrolment or severe hypertension according to WHO criteria or uncontrolled hypertension at the time of enrolment (systolic blood pressure ≥ 180 mm Hg)´
9. Previous chemotherapy for metastatic PCA.
10. Previous anti-hormonal treatment with abiraterone or any other investigational anti-hormonal treatment.
11. Cancer-related pain requiring opioid narcotics within 28 days before enrolment or an average pain score of > 3 on a visual analogue scale.
12. Presence of visceral metastases.
13. History of other malignancies other than PCA over the last 5 years (except basal cell carcinoma of the skin).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Phase I (Safety Lead-In): Occurrence of dose-limiting toxicity (DLT) during the first 4 weeks of treatment (after administration of 3 vaccinations and after a 1 week observation period | Up to 4 weeks
  Safety Lead in Portion:
  Patients will receive CV9104 at a starting dose of 1920 µg in weeks 1, 2 and 3. Safety lead-in patients will be observed for DLTs until 1 week after Vaccination 3 (week 4). In case no DLTs will be observed vaccinations will continue in weeks 5, 7, 9, 12, 15, 18 and 24, then every 6 weeks for up to 12 months after the first vaccination and then every 3 months thereafter until one of the criteria for study treatment discontinuation is met
Phase II (Randomised Portion): Overall Survival from time of randomisation- up to 3.5-4 years. | Overall survival will be assessed during the lifetime of the study

SECONDARY OUTCOMES:
Progression free survival from date of randomisation | Every 3 months for up to 2 years
Progression free survival from start of first subsequent systemic therapy | Every 6 months until 2 years
Percent change to maximal and to minimal PSA from baseline and before start of first subsequent systemic cancer therapy and from start of first systemic therapy to end of first subsequent systemic therapy | Every 3 months up to 2 years
Cellular and humoral immune response rate against the 6 antigens encoded by CV9104 | Immune responses will be assessed at baseline, in week 6 and week 24 after start of vaccination
Time to symptom progression based on FACT P score and subscores | Assessments at baseline, weeks 5, 9,18, 24 and every 3 months for up to 2 years
Absolute change and area under the curve from baseline EQ-5D score and pain sub-score | Assessments at baseline, weeks 5, 9,18, 24 and thereafter every 3 months for up to 2 years
Progression free survival from randomisation until second progression on first subsequent therapy | Every 3 and 6 months up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Stenzl, Prof. Dr., Principal Investigator — University Hospital of Tübingen; Dept. of Urology
Locations (48):
- Czechia (5):
  - Krajská zdravotní, a.s. - Nemocnice Chomutov, o.z.Onkologické oddělení, Chomutov
  - Fakultní nemocnice Olomouc, Urologická klinika, Olomouc
  - Multiscan, a.s, Oddělení klinické a radiační onkologie, Pardubice
  - Thomayerova nemocnice, Urologické oddělení, Prague
  - Krajská zdravotní, a.s. - Masarykova nemocnice Ústí nad Labem, Ústí nad Labem
- Institut Gustave Roussy, Villejuif, France
- Germany (16):
  - Universitätsklinikum Aachen Klinik für Urologie, Aachen
  - Vivantes Klinikum Am Urban Klinik für Urologie, Berlin
  - Medizinisches Zentrum Friedensplatz, Bonn
  - Universitätsklinikum Dresden Klinik und Poliklinik für Urologie, Dresden
  - Chirurgische Universitätsklinik Freiburg Klinik für Urologie, Freiburg im Breisgau
  - Urologikum Hamburg, Hamburg
  - Nationales Zentrum für Tumorerkrankungen Medizinische Onkologie, Heidelberg
  - Urologie am Nordplatz, Leipzig
  - UMM Universitätsmedizin Mannheim, Mannheim
  - Praxis Dr.schulze, Marklleeberg
  - Urologische Klinik und Poliklinik der Technischen Universität München Klinikum Rechts der Isar, Munich
  - Universitätsklinikum Münster Klinik und Poliklinik für Urologie, Münster
  - Studienpraxis für Urologie, Nürtingen
  - Ortenau Klinikum Urologie und Kinderurologie, Offenburg
  - Urologische Klinik Dr. Castingius München, Planegg
  - Universitätsklinik für Urologie, Tübingen
- Poland (8):
  - Medica Pro Familia Krakow, Krakow
  - Centrum Urologiczne Sp. z o.o., Mysłowice
  - Centralny Szpital Kliniczny MSWiA, Klinika Onkologii I Hematologii, Warsaw
  - Szpital Sw. Elżbiety - Mokotowskie Centrum Medyczne, Warsaw
  - Instytut M. Curie-Skłodowskiej Centrum Onkologii, Warsaw
  - NZOZ Magodent, Centrum Medyczne Ostrobramska, Oncologii Klinicznej i Chemíoterapii, Warsaw
  - Profesorskie Centrum Medyczne OPTIMUM Wrocław, Wroclaw
  - Szpital Uniwersytecki, Katedra i Klinika Urologii i Onkologii Urologicznej, Wroclaw
- Spain (5):
  - Hospital de Madrid Norte Sanchinarro Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - Hospital Clínico Virgen de la Victoria Campus Universitario de Teatinos s/n, Málaga
  - Clínica Universitaria de Navarra Departamento de Oncología, Pamplona
  - Complejo Hospitalario Universitario Santiago Departamento de Oncología, Santiago de Compostela
  - Instituto Valenciano de Oncología Unidad de Investigación Clínica, Valencia
- Sweden (5):
  - "Sahlgrenska Universitetssjukhuset Urologmottagningen, Gothenburg
  - Skånes Universitetssjukhus Malmö Urologmottagningen, Malmo
  - Universitetssjukhuset Örebro Urologmottagningen, Örebro
  - Karolinska Universitetssjukhuset Solna Urologiska kliniken, Stockholm
  - Akademiska sjukhuset Urologmottagningen, Uppsala
- Switzerland (4):
  - Universitätsspital Basel Medizinische Onkologie, Basel
  - Kantonsspital Graubünden Department Innere Medizin Hämatologie und Onkologie, Chur
  - CHUV Centre Pluridisciplinaire d'Oncologie, Lausanne
  - Kantonsspital St. Gallen Department Innere Medizin Hämatologie Medizinische Onkologie, Sankt Gallen
- United Kingdom (4):
  - Royal Free Hospital, London
  - Nottingham City Hospital Department of Oncology, Nottingham
  - Clatterbridge Cancer Centre, Wirral, Merseyside
  - York Hospital, York

REFERENCES:
- See also: Click here for more information about CureVac — http://www.curevac.de